CLINICAL TRIAL: NCT04534907
Title: Effectiveness of the Immersive Virtual Reality (VR) Treatment With Cognitive Behaviour Therapy (CBT) for Obsessive-Compulsive Disorder (OCD) : A Randomized Controlled Study
Brief Title: The Effect of Immersive Virtual Reality Treatment With Cognitive Behaviour Therapy for Obsessive-Compulsive Disorder
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Mental Health Center (Other)
Responsible Party: Principal Investigator, Zhen Wang, vice-president, Shanghai Mental Health Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SMHC-OCD-009
Record Dates: First submitted 2020-08-23; First posted 2020-09-01 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Obsessive-Compulsive Disorder; Virtual Reality
Keywords: Virtual Reality; cognitive-behavioral therapy; Exposure and Response /Ritual Prevention
MeSH Terms: conditions — Obsessive-Compulsive Disorder

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- VR(ERP） (Active Comparator): The combination of exposure and response prevention (ERP) and VR will be applied twice a week for the fist two weeks. For the next four weeks, this treatment will be applied once a week. 8 times in total
  Interventions: Combination Product: The combination of exposure and response prevention (ERP) and VR
- traditional ERP (Active Comparator): The traditional ERP will be applied twice a week for the fist two weeks. For the next four weeks, this treatment will be applied once a week. 8 times in total
  Interventions: Behavioral: Traditional ERP

INTERVENTIONS:
Combination Product: The combination of exposure and response prevention (ERP) and VR — The combination of exposure and response prevention (ERP) and VR aimed to investigate the combination of an immersive virtual reality environment (VRE) alongside therapist delivered CBT to reduce anxiety when the OCD patients were induced by virtual scene.Specially, patients will get the first CBT session in the first week for 90 minutes in order to gather detailed information of individual's symptom. Then the next 2 weeks, patients will get VR+ERP session twice a week. From the fourth week to the seventh week, patients weill get VR+ERP session once a week. In the end of the eighth week, patients will get the last session of the exposure-based CBT for relapse prevention.
  Arms: VR(ERP）
Behavioral: Traditional ERP — Patients will achieve the exposure based CBT for total 10 times excluding 8 sessions of ERP. Structured protocol described by Foa et al., 2012. Specially, patients will get the first CBT session in the first week for 90 minutes in order to gather detailed information of individual's symptom. Then the next 2 weeks, patients will get ERP session twice a week. From the fourth week to the seventh week, patients weill get ERP session once a week. In the end of the eighth week, patients will get the last session of the exposure-based CBT for relapse prevention.
  Arms: traditional ERP

SUMMARY:
This study will evaluate the clinical effectiveness ofthe Immersive Virtual Reality alongside exprosure and response Prevention (ERP) Treatment in cognitive-Behavioral Therapy for Obsessive-compulsive Disorder, and the underlying neural mechanism by electroencephalography (EEG) and eye-tracking methodology .

DETAILED DESCRIPTION:
The current study aims to the clinical effectiveness of the Immersive Virtual Reality alongside exprosure and response Prevention (ERP) Treatment in cognitive-Behavioral Therapy for Obsessive-compulsive Disorder. 30 OCD patients whose symptom were mainly associated with "contamination/clean" , "Symmetry/precision", "Examination" and "Sex" will be randomized into two groups (i.e. VR ERP or ERP). The treatment will be performed twice a week for the first two weeks. And for the next 4 week, the treatment for OCD patients will be undertook once a week. There will be 8 times in total. The investigators will assess thhe OCD patients'symptom severity in the baseline, 2 weeks, 4weeks and after 8 weeks of the whole combined treatment. Through the study, Yale-Brown Obsessive Compulsive Scale（Y-BOCS）, the Obsessive Compulsive Inventory-Revised (OCI-R), the Beck Depression Inventory (BDI), the Beck Anxiety Inventory (BAI), Perceived Stress Scale (PSS), Pittsburgh sleep quality index (PSQI) and side-effect questionnaire will be obtained by a trained investigator. The patients will also get individual's data of EEG and eye-movement.

ELIGIBILITY:
Inclusion Criteria:

* age: 18-50 years old;
* Diagnostic and Statistical Manual of Mental Disorders (DSM-5) criteria for OCD;
* Y-BOCS total score > or = 16, discontinued medication for at least 8 weeks before
* the enrollment or the paitients' clinical medication is stable for at least a month (the dose and the types of drugs) .>or＝9 years education

Exclusion Criteria:

* Any axis I psychiatric disorder comorbidity
* Participants who have received any forms of psychological therapy in the past.
* Patients cannot tolerate or adapt to the somatic discomfort caused by VR .
* Prior history of neurological disease (e.g., epilepsy) or brain surgery for traumatic brain injury
* Participants with claustrophobic, heart pacemaker, mechanical heart valve, mechanical implant such as an aneurysm clip, hip replacement, or any other pieces of metal that have accidentally entered their body.
* Any current significant medical condition.
* serious suicide risk

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Yale-Brown Obsessive Compulsive Scale(Y-BOCS) score | from baseline to 8weeks
  It assesses the severity of OCD symptoms. The Y-BOCS scale ranges from 0 to 40, with 0 being no symptoms and 40 being severe.The responder on Y-BOCS is defined as a Y-BOCS decrease at least 35% from the baseline at post-treatment.

SECONDARY OUTCOMES:
Change in Obsessive Compulsive Inventory-Revised(OCI-R) | from baseline to 8weeks
  It is an inventory of OCD symptoms with 18 items that are rated on a 5-point Likert scale. Total scores range from 0 to 72, with higher scores indicating more severe OCD symptoms.
Change in Beck Depression Inventory(BDI) | from baseline to 8weeks
  It consists of 21 items and uses a 0 to 3 severity scale. Total scores range from 0 to 63, with higher scores indicating more severe depression symptoms.
Change in Beck Anxiety Inventory (BAI) | from baseline to 8weeks
  It is an inventory of anxiety symptoms with 18 items that are rated on a 5-point Likert scale(0 to 4). Total scores range from 0 to 72, with higher scores indicating more severe anxiety symptoms.
Chinese version of Working Alliance Inventory-Short Form (WAI-SR) | assessed only once after the entire treatment at the end of the eighth week. (at the end week 8 )
  The WAI-SR measures three domains of the therapeutic alliance: (a) agreement between patient and therapist on the goals of the treatment (Goal); (b) agreement between patient and therapist about the tasks to achieve these goals (Task); and (c) the quality of the bond between the patient and therapist (Bond).
Simulator Sickness Questionnaire(SSQ) | The SSQ should be assessed each time after the VR+ERP treating for OCD patients. (at week 2, 3, 4, 5, 6, 7)
  The SSQ has been traditionally used for simulator motion sickness measurement,The SSQ was administered immediately after each task, and the order of work was determined using the Latin square design.

CONTACTS AND LOCATIONS:
Overall Officials: Zhen Wang, PhD,MD, Principal Investigator — Shanghai Mental Health Center
Locations (1):
- Shanghai Mental Health Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No